CLINICAL TRIAL: NCT02151708
Title: Efficacy of Motilitone on Gastric Emptying in Patients With Functional Dyspepsia:
Brief Title: Efficacy of Motilitone on Gastric Emptying in Patients With Functional Dyspepsia: Evaluation Using MRI Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Poong-Lyul Rhee, Clinical Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-12-026
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Dyspepsia
Keywords: accommodation, emptying,motilitone
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- motilitone 90mg (Active Comparator): Eligible subjects were randomly allocated in a 1:1:1 ratio to receive either 90mg motilitone or 180mg motilitone or placebo motilitone three times daily for 2weeks.
  Interventions: Drug: motilitone
- motilitone 180mg (Active Comparator): Eligible subjects were randomly allocated in a 1:1:1 ratio to receive either 90mg motilitone or 180mg motilitone or placebo motilitone three times daily for 2weeks.
  Interventions: Drug: motilitone
- placebo (Placebo Comparator): Eligible subjects were randomly allocated in a 1:1:1 ratio to receive either 90mg motilitone or 180mg motilitone or placebo motilitone three times daily for 2weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Eligible subjects were randomly allocated in a 1:1:1 ratio to receive either 90mg motilitone or 180mg motilitone or placebo motilitone three times daily for 2weeks.
  Arms: placebo
Drug: motilitone — Eligible subjects were randomly allocated in a 1:1:1 ratio to receive either 90mg motilitone or 180mg motilitone or placebo motilitone three times daily for 2weeks.
  Arms: motilitone 180mg; motilitone 90mg

SUMMARY:
Functional dyspepsia (FD) is a disorder characterized by chronic or recurrent upper abdominal pain or discomfort in the absence of a specific structural cause.1 Several mechanisms have been suggested to underlie dyspeptic symptoms. In a barostat study by Tack et al.2, impaired gastric accommodation to a meal was found in 40% of patients with FD, and this abnormality was associated with early satiety. Delayed gastric emptying (GE) was also found in almost 40% of patients with FD, and was associated with the symptoms of postprandial fullness, vomiting and early satiety.3-5 Improving gastric accommodation and prokinetic effect seem to be an attractive physiological target in patients with FD. Motilitone (Dong-A ST, Yongin, Korea) is a new herbal drug that was launched in December 2011 in Korea for treating patients with FD. It has multiple mechanisms of action such as fundus relaxation, visceral analgesia and prokinetic effects.6 The current study aims to evaluate effects of motilitone on gastric emptying and accommodation after a meal in patients with FD using three-dimensional gastric volume measurements by magnetic resonance imaging (MRI). Patients are randomly allocated to receive either motilitone 90 mg daily, motilitone 180 mg daily or placebo in a double blinded manner. After 2 weeks of treatment, patients undergo gastric MRI. The primary endpoint is gastric emptying rate. The secondary endpoints are gastric accommodation and symptom improvement.

DETAILED DESCRIPTION:
Same as above

ELIGIBILITY:
Inclusion Criteria:

1. 20 and 70 years of age
2. Diagnosed of functional dyspepsia patients by ROME III diagnostic criteria
3. Symptom scores three-point by 8 kinds of symptoms on NDI-K table
4. Signed written informed consent.

Exclusion Criteria:

1. Any functional GI diease
2. Previous abdominal surgery
3. pregnancy or lactation
4. Other conditions likely to interfere with study procedures. as judged by the investigator
5. Allergic history to motilitone
6. Contraindications to MRI
7. Significant cardiopulmonary disease
8. Significant renal(serum creatinine level≥1.5 x the upper normal limit) or liver (AST or ALT≥2.5xULN)disease
9. Can not be stopped taking medications that gastric motility booster and antacid prior to the start of the study
10. Uncontrollable diabetes mellitus (HbA1C>7%)
11. Any malignancies within 5 years prior to the start of the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation in gastric emptying rate after the test meal | Evaluation in gastric emptying rate 120min after the test meal

SECONDARY OUTCOMES:
The secondary endpoints are gastric accommodation and symptom improvement. | This outcome is measured on day 14 after 2 weeks of treatment
Change in total gastric volume (TGV) after the test meal | This outcome is measured on day 14 after 2 weeks of treatment.The change is defined as difference between TGV 15min after the test meal and at the pre-test meal.
Gastric emptying rate(GE) | GE 15min 30min 60min after the test meal.
Change in proximal total gastric volume (TGV) after the test meal | The chanfe is defined as difference between proximal TGV 15min after the test meal
Change in proximal to distal total gastric volume (TGV) ratio afrer the test meal | The change is defined as difference between proximal TGV 15min after the test meal and at the pre test meal

CONTACTS AND LOCATIONS:
Overall Officials: Poong-Lyul Rhee, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center,Sungkyunkwan University School of Medicine, Seoul, South Korea